CLINICAL TRIAL: NCT02767869
Title: Effect of Banaba (Lagerstroemia Speciosa) on Metabolic Syndrome, Insulin Secretion and Insulin Sensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, PHD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BANABA-MS
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic syndrome; central obesity; Banaba; insulin secretion; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Banaba (Experimental): Banaba capsules, 500mg, two times per day before meals during 90 days
  Interventions: Drug: Banaba
- Placebo (Placebo Comparator): Calcined magnesia capsules, 500mg, two times per day before meals during 90 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Banaba — Banaba capsules of 500 mg two times per day before meals with a total dosis of 1000 mg per day.
  Other Names: Lagerstroemia speciosa
  Arms: Banaba
Drug: placebo — Calcined magnesia capsule, 500 mg, two times per day before meals with a total dose per day of 1000 mg
  Other Names: calcined magnesia
  Arms: Placebo

SUMMARY:
The Metabolic Syndrome is a high prevalence disease worldwide. About a quarter of the adult population suffers the disease.

Banaba has shown evidence that has on metabolic syndrome, insulin sensitivity and insulin secretion.

The investigators hypothesis was that the the administration of resveratrol modifies the metabolic syndrome, insulin sensitivity and insulin secretion.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial was carried out in 24 patients with a diagnosis of metabolic syndrome in accordance with the International Diabetes Federation (IDF). Waist circumference, glucose, insulin levels, and lipid profile were evaluated after a 75 g of dextrose load.

12 received Banaba, 500 mg, two times per day (1000 mg) before meals during 3 months.

The remaining 12 patients received placebo with the same prescription.

Area Under the Curve of glucose and insulin was calculated as well as total insulin secretion (insulinogenic index), first-phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

This protocol was approved by a local ethics committee and written informed consent was obtained from all volunteers.

Results are presented as mean and standard deviation. Intra and inter group differences were tested using the Wilcoxon signed-rank and Mann-Whitney U-test respectively; p≤0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes,
* Age between 30 and 60 years,
* Metabolic Syndrome according to the IDF criteria
* Waist circumference
* Man ≥90 cm
* Woman ≥80 cm

And two of the following criteria:

* High density lipoprotein
* Man ≤40 mg/dL
* Woman ≤50 mg/dL
* Fasting glucose ≥100 mg/dL
* Triglycerides ≥150 mg/dL
* Blood pressure ≥130/85 mmHg
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to resveratrol
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Previous treatment for the metabolic syndrome components
* Body Mass Index ≥39.9 kg/m2
* Fasting glucose ≥126 mg/dL
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Low density lipoprotein (c-LDL) ≥190 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Intstituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Lopez-Murillo LD, Gonzalez-Ortiz M, Martinez-Abundis E, Cortez-Navarrete M, Perez-Rubio KG. Effect of Banaba (Lagerstroemia speciosa) on Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion. J Med Food. 2022 Feb;25(2):177-182. doi: 10.1089/jmf.2021.0039. Epub 2021 Nov 2. PMID 34726501

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Banaba | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sample size was calculated in accordance of Jeyaseelan's clinical trial formula with a statistical confidence of 95%, statistical power of 80%, obtaining a total of 12 patients per group including 20% of expected loss.
Groups:
- Total: Total of all reporting groups
Arm/Group | Banaba | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (9.1) | 45.5 (6.5) | 45 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Body weight [Mean (Standard Deviation); unit: kg] — Body weight was evaluated through a bioimpedance digital scale and results are reported in kg with a decimal.
  kg | 76.5 (11.6) | 78.8 (10.3) | 77.6 (10.9)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (2.6) | 28.6 (3.8) | 28.6 (3.2)
Waist circumference [Mean (Standard Deviation); unit: cm] — Waist circumference was measured with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 97.0 (7.8) | 97.4 (8.8) | 97.2 (8.3)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Measure Description: Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP). The value was expressed on mmHg
  mmHg | 121.5 (12.9) | 122.6 (9.6) | 122.0 (11.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Measure Description: Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP). The value was expressed on mmHg
  mmHg | 76.5 (9.6) | 81.7 (5.5) | 79.1 (7.5)
Glucose 0' [Mean (Standard Deviation); unit: mg/dL] — Measure Description: The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 0 and 120 after a 75 g oral dextrose load.
  mg/dL | 106.9 (7.9) | 106.7 (6.6) | 106.8 (7.2)
Glucose 120' [Mean (Standard Deviation); unit: mg/dL] — Measure Description: The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal and at the minutes 30, 60, 90 and 120 after a 75 g oral dextrose load.
  mg/dL | 131.3 (27.2) | 138.3 (28.2) | 134.8 (55.4)
Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Measure Description: The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots to determine cholesterol
  mg/dL | 217.5 (48.3) | 197.7 (37.3) | 207.6 (42.8)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Measure Description: The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine triglycerides
  mg/dL | 204.4 (38.9) | 200.8 (80.6) | 202.6 (59.75)
High-density lipoprotein-cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into aliquots: the first was immediately analyzed to determine high-density lipoprotein-cholesterol (HDL-C)
  mg/dL | 60.8 (18.1) | 57.3 (20.4) | 59.0 (19.2)
Low-density lipoprotein-cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood was centrifuged at 2000 rpm and serum was separated into two aliquots: the first was immediately analyzed to determine low-density lipoprotein-cholesterol (LDL-C).
  mg/dL | 108.1 (39.3) | 108.0 (35.3) | 108.0 (37.3)
Area under the curve (AUC) glucose [Mean (Standard Deviation); unit: mg*min/dL] — The area under the curve (AUC) of glucose, (0.5 * glucose (G) 0´ + (G 30´+G 60´ + G 90´) + 0.5 * G 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperglycemia.
  mg*min/dL | 18567.6 (3480.6) | 19336.3 (3224.7) | 18951.9 (3352.6)
Area under the curve (AUC) insulin [Mean (Standard Deviation); unit: uU*min/mL] — The area under the curve (AUC) of insulin, (0.5 * Insulin (I) 0´ + (I 30´+I 60´ + I 90´) + 0.5 * I 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperinsulinemia.
  uU*min/mL | 8445.9 (2384.8) | 7669.7 (2109.5) | 8057.8 (2247.1)
Very low-density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mg/dL] | 41.0 (8.0) | 40.1 (7.7) | 40.5 (7.8)
Total insulin secretion [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion at baseline.
  index | 0.4 (0.2) | 0.4 (0.1) | 0.4 (0.1)
First phase of insulin secretion [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the frst phase of insulin secretion at baseline.
  index | 954.3 (285.3) | 910.3 (514.1) | 932.3 (399.7)
Insulin sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes.
  Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity at baseline
  index | 5.2 (1.4) | 5.1 (2.7) | 5.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Triglyceride Levels at Week 12
Description: The triglycerides will be evaluated at week 12 with enzymatic-colorimetric techniques.
Time Frame: Week 12
Population: All participants, including those who dropped out before the end were taken into account for statistical analysis (intention to treat)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 148.0 (43.0) | 199.9 (101.9)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney)

2. Primary Outcome: High Density Lipoprotein-cholesterol (HDL-C) Levels at Week 12
Description: The HDL-C levels will be evaluated at week 12 with enzymatic/colorimetric techniques.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 56.4 (11.2) | 58.4 (16)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.530, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Fasting Glucose Levels at Week 12
Description: The fasting glucose levels were evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 103.2 (7.4) | 104.2 (8.9)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.034, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Systolic Blood Pressure at Week 12.
Description: The systolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the systolic blood pressure at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 116.3 (9.8) | 122.6 (13.1)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney)

5. Primary Outcome: First Phase of Insulin Secretion at Week 12
Description: Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the frst phase of insulin secretion at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
index | 913.9 (490.3) | 651.0 (405.2)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.799, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Total Insulin Secretion at Week 12.
Description: Measure Description: The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
index | 0.3 (0.2) | 0.3 (0.1)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Total Insulin Sensitivity at Week 12
Description: Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
index | 5.1 (3.2) | 5.5 (2.3)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.878, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Waist Circumference at Week 12
Description: Waist circumference will be evaluated at baseline and at week 12 with a flexible tape
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
cm | 95.7 (7.9) | 97.0 (7.8)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.919, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Diastolic Blood Pressure at Week 12
Description: The diastolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the diastolic blood pressure at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 72.5 (9.2) | 76.5 (9.6)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.254, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Weight at Week 12
Description: The weight was measured at baseline and week 12 with a bioimpedance balance and the entered values reflect the weight at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
kg | 72.6 (8.6) | 72.2 (8.1)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.347, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Body Mass Index at Week 12
Description: The Body Mass index was calculated at baseline and at week 12 with the Quetelet index and the entered values reflect the body mass index at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
kg/m^2 | 28.4 (2.7) | 28.9 (5.7)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.227, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Total Cholesterol at Week 12
Description: The total cholesterol was estimated by standardized techniques at baseline and week 12 and the entered values reflect the total cholesterol level at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 210.0 (39.6) | 201.7 (34.8)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.410, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Low-density Lipoprotein-cholesterol (LDL-C) at Week 12
Description: The LDL-C levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the c-LDL levels at week 12
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Banaba | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL | 29.0 (8.0) | 39.9 (20.3)
Statistical Analysis 1: Comparison: Banaba vs Placebo; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 12-week study.
Arm/Group | Banaba | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Banaba (N=12) | Placebo (N=12)
softening of stool (Gastrointestinal disorders) | 9 (9) | 0 (0)
abdominal colic (Gastrointestinal disorders) | 3 (3) | 2 (2)
flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
abdominal swelling (Gastrointestinal disorders) | 1 (1) | 4 (4)
pyrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No